CLINICAL TRIAL: NCT06748742
Title: A Randomized Controlled Trial to Improve the Therapeutic Effect of Robot-assisted Radical Prostatectomy (RARP) Using Indocyanine Green Fluorescence Imaging
Acronym: ICG-RARP
Status: Active, not recruiting | Type: Observational
Sponsor: Liu Cheng (Other)
Responsible Party: Sponsor-Investigator, Liu Cheng, Chef Doctor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: ICG-RARP
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Prostate CA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Patients who underwent radical resection of prostate malignant tumor with anterior approach at Shanghai First People's Hospital
- Experiment Group: Patients who used ICG to identify and separate the bladder neck during anterior robot-assisted radical prostatectomy
  Interventions: Drug: In robot-assisted radical prostatectomy, indocyanine green fluorescent solution is injected through the urethra, and the position and structure of the urethra are observed by the device

INTERVENTIONS:
Drug: In robot-assisted radical prostatectomy, indocyanine green fluorescent solution is injected through the urethra, and the position and structure of the urethra are observed by the device — In robot-assisted radical prostatectomy, indocyanine green fluorescent solution is injected through the urethra, and the position and structure of the urethra are observed by using the fluorescence imaging equipment that comes with the device. Guided by real-time fluorescence imaging, the urethra is precisely dissected and severed in front of the bladder neck. Through this improved operation, the bladder neck is protected, the neck injury that is common in conventional surgical operations is reduced, and the reconstructive surgical operations necessary after loss are reduced, and the surgical efficiency is improved. By protecting the bladder neck, the sphincter is better preserved, postoperative urinary incontinence is reduced, and the surgical outcome is improved.
  Groups: Experiment Group

SUMMARY:
In Robotic Assistant Radical Prostatectomy (RARP), indocyanine green fluorescent solution is injected through the urethra, and the position and structure of the urethra are observed using the fluorescence imaging equipment that comes with the device. Guided by real-time fluorescence imaging, the urethra is precisely dissected and severed in front of the bladder neck. Through this improved operation, the bladder neck is protected, the neck injury that is common in conventional surgical operations is reduced, and the reconstructive surgical operations necessary after loss are reduced, and the surgical efficiency is improved. By protecting the bladder neck, the sphincter is better preserved, postoperative urinary incontinence is reduced, and the surgical outcome is improved

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with prostate cancer who underwent robot-assisted radical prostatectomy at Shanghai First People's Hospital Patients with naïve localized prostate cancer or locally advanced prostate cancer The patient > 18 years and < 85 years Before the surgery, the prostate MR scan sagittal view of the prostate in our hospital measured the separation of the bladder neck < 1cm The patient underwent robot-assisted laparoscopic radical resection of the prostate malignancy in our hospital with anterior approach The patient returned to normal after surgery, and there were no postoperative complications such as intestinal obstruction that affected the patient's blood routine and biochemical indicators

Exclusion Criteria:

Patients with metastatic prostate cancer Patients without preoperative puncture pathology Patients with sagittal bladder neck separation ≥ 1cm of prostate MR non-contrast prostate in our hospital before surgery Patients with preoperative examinations confirming that the enlarged prostate protrudes into the bladder floor Patients with preoperative examination confirming that the lesion is located at the tip of the prostate and near the bladder neck Patients with tumor stage reaching cT4 stage and possible invasion of bladder neck Patients who have undergone adjuvant therapy such as endocrine therapy and radiotherapy before surgery Patients with a history of any prostate surgery other than needle biopsy prior to radical resection of prostate malignancy Patients who have undergone resection of transurethral bladder lesions Patients who have undergone abdominal/pelvic surgery that makes it difficult to separate the prostate and surrounding structures during RARP Patients undergoing extended pelvic lymph node dissection during surgery Patients with posterior approach during surgery Patients with poor urinary continence due to any non-surgical factors after surgery Patients with a history of ICG allergy

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet all the inclusion criteria and have no exclusion criteria for any of the conditions
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The study subjects completed the follow-up results of 6 months after RARP | One month, three months, six months after surgery
  The resection margins of the postoperative pathology of the patients included in the study and the urinary continence at one, three, and six months follow-up after surgery; Repeat PSA values (to reflect the presence or absence of biochemical recurrence)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China